CLINICAL TRIAL: NCT03386604
Title: Physical Capacity of Patients With Chronic Obstructive Pulmonary Disease in Pulmonary Rehabilitation With and Without Supplementation of Whey
Brief Title: Physical Capacity of Patients With Chronic Obstructive Pulmonary Disease With and Without Supplementation of Whey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 72793717.0.0000.5327
Record Dates: First submitted 2017-12-05; First posted 2017-12-29 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Dietary Supplements; Rehabilitation
Keywords: Whey Protein
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Whey Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey protein + Rehabilitation (Experimental): Pulmonary rehabilitation will last 8 weeks covering 3 weekly sessions of supervised exercise and a weekly educational session. Patients will receive whey protein and will be instructed to take it daily for breakfast, diluted in milk or water (if they do not drink milk).
  Interventions: Dietary Supplement: Whey protein
- Placebo + Rehabilitation (Placebo Comparator): Pulmonary rehabilitation will last 8 weeks covering 3 weekly sessions of supervised exercise and a weekly educational session. Patients will receive placebo (maltodextrin) and will be instructed to take it daily for breakfast, diluted in milk or water (if they do not drink milk).
  Interventions: Dietary Supplement: Maltodextrin
- Control (No Intervention): Patients without pulmonary rehabilitation nor whey protein supplementation.

INTERVENTIONS:
Dietary Supplement: Whey protein — whey protein 40 g: energy value 160 kcal; carbohydrate 10 g; 25g proteins; total fat 2.3g; saturated fats 1.1 g; trans fat 0 g; dietary fiber 0 g; sodium 157 mg; calcium 264 mg.
  Arms: Whey protein + Rehabilitation
Dietary Supplement: Maltodextrin — Maltodextrin energy value 160 kcal.
  Arms: Placebo + Rehabilitation

SUMMARY:
Chronic obstructive pulmonary disease is characterized by obstruction to pulmonary airflow and dyspnea. These characteristics are a consequence of exposure to harmful gases and particles that lead to oxidative stress in the lungs together with an exaggerated inflammatory response. In addition to respiratory impairment, chronic obstructive pulmonary disease has systemic manifestations, nutritional alterations, and exercise limitation. Pulmonary rehabilitation is one of the most effective interventions in the treatment of chronic obstructive pulmonary disease, with one goal being to improve patient capacity. Whey protein supplementation, concomitant with physical activity for patients with chronic obstructive pulmonary disease, aims to stimulate protein synthesis and decrease muscle catabolism that may be caused by exercise. The investigators aimed to evaluate the effects of whey protein supplementation supplementation on the physical capacity, body composition and tissue functionality of patients with chronic obstructive pulmonary disease in a pulmonary rehabilitation program.

DETAILED DESCRIPTION:
A randomized clinical study will be carried out with 62 patients (31 patients per group) with chronic obstructive pulmonary disease who came from specialized departments of the Pulmonology Service of the Hospital de Clínicas of Porto Alegre and were referred to the pulmonary rehabilitation program of this institution. Patients will be evaluated in relation to anthropometry, body composition, blood biochemistry, phase angle, dietary intake, physical capacity, muscle strength and lung function. The data will be processed in the statistical program SPSS version 17.0 and for statistical analysis they will be tested for their normality by the Kolmogorov-Smirnoff test and after this definition will be applied specific tests for parametric or non-parametric data, being they presented in the form of mean and standard deviation or median, minimum and maximum, according to their distribution. The differences will be considered significant for values of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have been referred for pulmonary rehabilitation for chronic obstructive pulmonary disease diagnosis;
* Stable for the last 3 months and have no contraindications to exercise (no infection, acute myocardial infarction, malignant neoplasms, renal or hepatic disease, ascites / edema or neuromuscular disease);
* Be 40 years or older;
* Being literate;

Exclusion Criteria:

* Being a vegetarian;
* Make use of continuous oxygen;
* Present cognitive or functional changes that limit the execution of any of the proposed tests.
* Body mass index <21.0 kg / m² and ≥ 35.0 kg / m².

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Physical capacity through the maximum distance traveled | 8 weeks
  The test will be performed during 6 minutes on a previously measured surface with a distance of 30m, without additional oxygen support.

SECONDARY OUTCOMES:
Muscle strength through manual grip strength of dominant and non-dominant limbs | 8 weeks
  Measurement of grip strength with dynamometer is performed with the patient sitting comfortably, with the shoulder attached, the elbow flexed at 90º, the forearm in the neutral position and the cuff should be between 0 (zero) and 30º of extension, and should perform the greatest gripping force possible. Six measurements will be performed with a 15-second interval, alternating the hands, starting with the dominant upper limb.
Body composition (amount of muscle mass) wiht absorptiometry by dual emission of X-ray | 8 weeks
  The measurements will be obtained with the patient in the supine position, positioned in the area of equipment scanning, so that the sagittal line demarcated in this area passes under the center of some anatomical points such as the skull, spine, pelvis and legs, and without metal objects attached to the body.
Tissue functionality through phase angle | 8 weeks
  The evaluation of the phase angle will be performed by means of the electric bioimpedance apparatus. The measurements will be obtained with the patient in dorsal decubitus, barefoot, with the lower limbs slightly apart and without metal objects attached to the body, with electrodes placed on the right hand and foot. Diuretic medications should be stopped 24 hours before the test, physical activities should be avoided until 8 hours before and a 4 hour fast will be requested.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina G De Souza, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided